CLINICAL TRIAL: NCT03221348
Title: A Phase I Open-label, Multiple Dose Study of CHO-H01 Administered Intravenously as a Single Agent to Subjects With Refractory or Relapsed Follicular Lymphoma
Brief Title: A Phase I Study of Intravenous CHO-H01 in Patients With Refractory or Relapsed Follicular Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cho Pharma Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FOLHAT-001
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: 3+3 sequential cohort design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label treatment (Experimental): Study drug (CHO-H01) administered on Day 1 of 28 day cycles up to 6 cycles total.
  Interventions: Biological: CHO-H01

INTERVENTIONS:
Biological: CHO-H01 — Glyco-engineered anti-CD20 antibody

SUMMARY:
This is a single-arm open label trial to explore the tolerability, safety, PK, PD, and anti-tumor activity of various doses and schedules of CHO-H01 administered as monotherapy in subjects with follicular lymphoma.

Groups of 6 subjects are planned for each cohort. The first 3 patients of each cohort will be evaluated to determine if it is appropriate to proceed with the additional 3 patients at that dose and schedule.

DETAILED DESCRIPTION:
This is a single-arm open label trial to explore the tolerability, safety, PK, PD, and anti-tumor activity of various doses and schedules of CHO-H01 administered as monotherapy in subjects with follicular lymphoma. This is not an MTD study, but an evaluation of optimum biological activity.

Groups of 6 subjects are planned for each cohort. The first 3 patients of each cohort will be evaluated to determine if it is appropriate to proceed with the additional 3 patients at that dose and schedule.

Schema 1:

1 mg/kg administered on D1 of Cycle 1 and D1 of subsequent 28 day cycles. Up to 6 cycles total are planned per subject.

Schema 2-3 Details to be determined after analysis of first 3-6 patients treated on Schema 1. Doses may be either escalated or de-escalated, or modified for Cycles 2-6 relative to Cycle 1. Schedules to be explored could include multiple doses with the first cycle: D1, D8 of 28 day cycles and D1, D8, D15 of 28 days cycles. In no case will individual doses exceed 10mg/kg.

Decisions on whether to proceed with a schema and details of selected dose and schedule will be made during cohort data review meetings by a Clinical-Scientific Review Team (CSRT) comprised of the trial investigators and Medical/Clinical and Safety representatives from the Sponsor. Ad hoc members will be consulted as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years Histologically confirmed, measurable, CD20 positive Follicular B cell lymphoma with an indication for treatment for which there is no therapy of curative potential or of higher priority
* Life expectancy of greater than 1 year
* ECOG performance status of 0 to 1
* Last dose of prior anti-cancer therapy must be at least 56 days (or two half-lives for proteins, whichever is greater) prior to the first administration of the study drug (to satisfy the recognized requirement of at least 5 times the terminal half-life period for most drugs currently used, including most receptor tyrosine kinase (RTK) inhibitors).
* Acute toxicities from any prior therapy, surgery, or radiotherapy must have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade 0 or 1.
* Subject must be willing and able to provide fresh tumor at Screening. Subjects will be asked to provide additional needle biopsy samples on C2D8 and C4D8. Archival tumor biopsy (i.e., tissue block or series of ≈10 slides) is requested if available, and should be provided during the Screening period.
* Local laboratories may be used for standard laboratory assessments:

Adequate bone marrow function defined by: absolute neutrophil count (ANC) of ≥ 1.5 x 109/L, platelet count of ≥ 100.0 x 109/L, and hemoglobin ≥9.0 g/dL.

Adequate hepatic function defined by: serum total bilirubin < 2 mg/dl (unless resulting from hemolysis), aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x ULN (or ≤ 5 x ULN in subjects with liver metastases).

Adequate renal function assessed by: serum creatinine within normal limits, or creatinine clearance (by Cockcroft Gault formula) ≥ 50 mL/min for subjects in whom serum creatinine may not adequately reflect renal function.

* Must have measurable disease as described in Lugano Revised Criteria for Response. This assessment is the responsibility of the investigator who may use local radiology to support this assessment.
* Willing and able to understand and sign an informed consent form and to comply with all aspects of the protocol.
* Willingness to use effective methods of contraception.
* Adequate T cell immune parameters - CD4 >500/mcL, CD8 > 250/mcL
* Bone marrow biopsy revealing adequate hematologic reserves

Exclusion Criteria:

* Evidence of circulating tumor cells >500 cells/microliter of lymphocytes or equivalent
* History of allergic reactions to any component of the study drug
* Autoimmune disease (Exceptions: autoimmune thyroiditis)
* Concomitant use of systemic corticosteroids
* History of seizure disorder
* History of Central Nervous System (CNS) metastases or seizure disorder related to the malignancy.
* History of symptomatic congestive heart failure (CHF), unstable angina pectoris, unstable atrial fibrillation; cardiac arrhythmia
* Non-manageable electrolyte imbalances, including hypokalemia, hypocalcemia, hypomagnesemia, and hypomagnesemia, of Grade 2 or greater (NCI-CTCAE v. 4.0)
* Any uncontrolled intercurrent illness, infection, or other condition that could limit study compliance or interfere with assessments
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Adverse drug reactions | 28 days
  Treatment-emergent adverse events and clinically significant laboratory values assessed for each subject and aggregated by type, frequency and severity by treatment cohort
Pharmacodynamic assessment of Immune cell activation | 64 days
  Gene expression of immune cell activation following treatment compared to baseline

SECONDARY OUTCOMES:
Clinical response | 8 weeks
  Lugano Revised Criteria for Response
Serum drug concentration | 72 hours
  Serum drug concentration measured at different times following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dahl, PhD, Study Director — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: No